CLINICAL TRIAL: NCT05088915
Title: Adolescent BREATHE Primary Care Intervention for PTSD (PCIP) Randomized Feasibility Trial
Brief Title: Adolescent PCIP Randomized Feasibility Trial
Acronym: APCIP
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Addressing potential changes to study setting.
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Lauren Ng, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-000207
Record Dates: First submitted 2021-09-29; First posted 2021-10-22 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Post-Traumatic Stress Disorder in Adolescence; Post Traumatic Stress Disorder
Keywords: Adolescent; Primary Care; PTSD; Post Traumatic Stress Disorder; Randomized Feasibility Trial; TF-CBT
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This study will utilize a hybrid effectiveness-implementation approach to conduct a randomized pilot feasibility trial of the PCIP screening and intervention protocol in adolescent primary care with two treatment arms:
  1. PCIP delivered through telehealth (computer or smartphone delivered videocall)
  2. Treatment as usual (TAU)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BREATHE Primary Care Intervention for PTSD (PCIP) (Experimental): BREATHE PCIP is a treatment for Post-Traumatic Stress Disorder (PTSD) symptoms for use with individuals who have a diagnosis of PTSD or "probable PTSD." The treatment will be considered delivered when patients have learned and practiced breathing retraining and have discussed the symptoms of PTSD (Sessions 1 through 3).
  Interventions: Behavioral: Primary Care Intervention for PTSD (PCIP)
- Treatment As Usual (Active Comparator): Receive standard care treatment and provided information on free or low cost mental health care referrals in the Los Angeles Area.
  Interventions: Behavioral: Treatment As Usual

INTERVENTIONS:
Behavioral: Primary Care Intervention for PTSD (PCIP) — This program is adapted from the "B.R.E.A.T.H.E. - Brief Relaxation, Education and Trauma Healing: A Brief Intervention for Persons with PTSD and Co- Occurring Serious Mental Health Conditions. Treatment Program Manual and Patient Handouts (Version 3) by Kim T. Mueser, Rachael Fite, Stanley D. Rosenberg, and Jennifer D. Gottlieb.
  Other Names: PCIP
  Arms: BREATHE Primary Care Intervention for PTSD (PCIP)
Behavioral: Treatment As Usual — Receive standard care treatment and are provided information on free or low cost mental health care referrals in the Los Angeles Area.
  Arms: Treatment As Usual

SUMMARY:
There are three research questions: (1) whether the Primary Care Intervention for PTSD (PCIP) improves health outcomes; (2) whether and how the PCIP can be sustainably delivered via telehealth; and (3) how PCIP compares to treatment as usual (TAU) participants.

The mixed methods randomized feasibility trial of the protocol will be measured by the RE-AIM framework (Reach, Effectiveness, Adoption, Implementation, Maintenance) (n=44 patients and their care givers). We will collect data on patient, caregiver, and clinic staff participation, retention, and satisfaction (Reach and Adoption), change in hypothesized treatment mechanisms and symptoms (Effectiveness), and facilitators and barriers to intervention delivery and fidelity (Implementation). We will,

1. Assess the reach and adoption of the protocol by analyzing quantitative data on patient and clinic staff participation, retention, and satisfaction;
2. Explore the effectiveness of the protocol through medical record review, quantitative assessments at baseline and post-treatment, and semi-structured qualitative interviews at baseline and post-treatment to:
3. Evaluate the implementation of the screening and intervention protocol with post-intervention semi-structured qualitative interviews to assess facilitators and barriers to intervention delivery, quantitative fidelity scales, observation of screening, and review of intervention audio recordings to assess fidelity to the protocol and intervention process.

ELIGIBILITY:
Inclusion Criteria:

1. Patient referred to the SHARK Program
2. Patients must be at least 12 years old
3. Screened for probable PTSD on UCLA RI, or at provider discretion of clinical relevancy.
4. If patient is under 18 years old, the patient's legal guardian is able and willing to provide informed consent for the patient to participate in the study;
5. Patient is able to complete study activities in English.

Exclusion Criteria:

1. Suicidal ideation with a plan within the last two weeks or a suicide attempt within the past 30 days;
2. Inability to provide informed consent or assent, and/or complete procedures in English.

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD Knowledge | Day 0 baseline, 10 months
  Changes in levels of PTSD Knowledge measured by the PTSD Knowledge Test (0-14, higher scores indicating more PTSD knowledge)
Change in Trauma-Related Cognitions | Day 0 baseline, 10 months
  Changes in post-traumatic cognitions measured by the Post-Traumatic Cognitions Inventory (1-7, Higher scores indicating more post traumatic cognitions)
Change in Self-Reported Arousal | Day 0 baseline, 10 months
  Changes in PTSD related arousal levels measured by the Composite Autonomic Symptom Score (COMPASS-31; 0-100 total, Higher scores indicating higher arousal)
Change in Stress Management Skill Use | Day 0 baseline, 10 months
  Changes in PTSD related arousal levels measured Measure of Adolescent Coping Strategies (MACS; Total 0-102, higher scores indicate higher use of specified coping), and use of the breathing retraining techniques as measured by self-reports during in-session review.
Intervention Implementation and Acceptability | Day 0 baseline, 10 months
  Qualitative interviews will include questions regarding acceptability of treatment including treatment via telehealth. Additionally, data will be collected regarding participant completion of therapy, no show rates, barriers to treatment, and attendance. Additionally, study therapists will complete qualitative and quantitative measures regarding intervention delivery feasibility and study protocols.

SECONDARY OUTCOMES:
Change in PTSD Symptoms | Day 0 baseline, 10 months
  Changes in PTSD related symptoms measured by the UCLA Child/Adolescent PTSD Reaction Index for DSM-5 Brief Screen (total 0-44; Higher scores indicate higher likelihood of PTSD and symptom-related distress and impairment)
Change in Trauma Symptoms | Day 0 baseline, 10 months
  Changes in trauma related symptoms measured by The Child PTSD Symptom Scale (CPSS-5-SR) Self Report (total 0-80, Higher scores indicated greater symptom severity).
Change in Adverse Childhood Experiences | Day 0 baseline, 10 months
  Changes in Adverse Childhood Experiences measured by the Pediatric ACEs and Related Life Events Screener (PEARLS; 0-19, higher scores indicate higher risk of traumatic stress.
Change in Depression Symptoms | Day 0 baseline, 10 months
  Changes in depression symptoms measured by the Center for Epidemiologic Studies Depression Scale (CES-DC) Self Report (total 0-60, Higher scores indicate higher symptom severity).
Change in Depression Symptoms | Day 0 baseline, 10 months
  Changes in depression symptoms measured by the Patient Health Questionnaire (PHQ-9;0-27; Higher scores indicate higher symptoms and likelihood of depression)
Change in Anxiety Symptoms | Day 0 baseline, 10 months
  Changes in anxiety symptoms measured by the Revised Children's Anxiety and Depression Scale (RCADS) Self Report (total 0-141, Higher scores indicating higher symptom severity).
Change in Functional Impairment | Day 0 baseline, 10 months
  Changes in functional impairment measured by The Columbia Impairment Scale (C.I.S.; 0-52, Higher scores indicate greater impairment).
Change in pro-inflammatory cytokine biomarkers | Day 0 baseline, 10 months
  Changes in pro-inflammatory cytokines including TNF-α, IL-6, IFN-γ and IL-1ß will be analyzed from Dried Blood Spots (DBS)
Change in pro-inflammatory transcription factor activation | Day 0 baseline, 10 months
  Changes in pro-inflammatory transcription factor activation including NF-κB/Rel will be analyzed from Dried Blood Spots (DBS)
Change in Substance Use | Day 0 baseline, 10 months
  Changes in substance use and misuse measured by CRAFFT Adolescent Substance Use Screen (0-9, Higher scores indicate higher risk for substance misuse)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren C Ng, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No